CLINICAL TRIAL: NCT03864783
Title: The Effect of Curcumin on Liver Fat Content in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-18045227
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Insulin Resistance; Glucose Tolerance Impaired; Obesity, Abdominal
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Glucose Intolerance; Obesity, Abdominal | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: At the end of the randomization visit, the patients will randomly be assigned to one of two interventions: 6 weeks of Meriva® (two capsules of 500 mg (corresponding to 200 mg curcumin) twice daily) or identically looking placebo (two capsules twice daily). There will be a stratification with respect to HbA1c, ensuring that if we include people with HbA1c ≥ 48 mmol/mol, they will be equally distributed in the two treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The supplier of Meriva® and placebo capsules (Indena® Aps, Milan, Italy) sends the tablets to the research department. After packaging of tablets in bags with tablets for 42 days (+7 extra tablets) and labelling of bags with a "bag number", a person not otherwise involved in the study will generate a list with a randomization number and a "bag number" using a random list generator. When an investigator enrols a participant in the study, the participant is assigned with a randomization number (in consecutive order), and the corresponding "bag number" will be handed to the participant. An emergency code will be kept at Gentofte Hospital. If a subject develops adverse events (AEs) that demand knowledge of the content of the intervention, the code may be broken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Meriva®) (Experimental): Meriva® 500 mg tablet (contains 100 mg curcumin) Dosage: 2 tablets twice daily for 42 days (+/- 3 days)
  Interventions: Dietary Supplement: Curcumin (Meriva®)
- Placebo (Placebo Comparator): Placebo. Dosage: 2 tablets twice daily to mimic Meriva® tablets.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Dietary Supplement: Curcumin (Meriva®) — Experimental drug:
  Meriva® 500 mg tablet (contains 1 mg curcumin)
  Arms: Curcumin (Meriva®)
Drug: Placebo Oral Tablet — Placebo:
  Contains same ingredients as Meriva®, apart from curcumin. Similar in appearance to Meriva®.
  Arms: Placebo

SUMMARY:
The majority of obese have non-alcoholic fatty liver disease (NALFD). Currently, no pharmacological agents are licenced for the prevention or treatment of NAFLD, and weight loss, notoriously difficult to obtain (and specially to maintain), remains the only treatment option. Interestingly, curcumin, a phenolic compound extracted from the turmeric root, has from in vitro and animal studies shown promising effects in preventing and treating NAFLD, and the sparse available human data point in the same direction; but solid human data are missing. This study will delineate the effects of curcumin when treating NAFLD in humans.

The primary aim of this study is to investigate the effect of 6 weeks of curcumin on liver fat content (assessed by magnetic resonance spectroscopy (MRS)) in obese subject with NAFLD. Additionally, a range of secondary endpoints have been chosen in order to delineate the role of NAFLD in the newly discovered liver-alpha cell axis governing circulating levels of the glucose-mobilising pancreatic alpha cell hormone glucagon and, thus, to elucidate the link between liver fat content and the risk of developing reduced glucose tolerance and type 2 diabetes (T2D). Also, the anti-inflammatory effect of curcumin will be elucidated, as inflammatory markers will be measured before and after intervention. Furthermore, the effect of curcumin will be measured by measuring the following parameters before and after intervention: Transient elastography, anthropometric measurements, body weight, appetite, food-consumption, calory balance, resting energy expenditure, gut microbiota, bioimpedance measures, visceral- and subcutaneous fat, glucose tolerance, lipids, blood pressure, pulse, liver parameters (blood-tests) and adipokines. During the oral glucose tolerance test before and after intervention, incretin hormones, glucagon, amino acids, insulin, c-peptide and urea will be measured.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing worldwide. Obesity and its associated complications represent an enormous burden for obese individuals, their families, healthcare systems and societies. Non-alcoholic fatty liver disease (NAFLD) has emerged as a frequent and serious complication of obesity. Steatosis, the benign and potentially reversible form of NAFLD, may progress to a more severe form, non-alcoholic steatohepatitis (NASH), which can result in fibrosis and ultimately liver cirrhosis, and rarely hepatocellular carcinoma. The majority of obese have NAFLD. Currently, no pharmacological agents are licenced for the prevention or treatment of NAFLD, and weight loss, notoriously difficult to obtain (and specially to maintain), remains the only treatment option. Interestingly, curcumin, a phenolic compound extracted from the turmeric root, has from in vitro and animal studies shown promising effects in preventing and treating NAFLD, and the sparse available human data point in the same direction; but solid human data are missing. This study seeks to investigate the effects of curcumin on treating NAFLD in humans by looking at the effects of ingestion of curcumin for 6 weeks in obese subject with NAFLD on lipid, glucose and protein metabolism.

In this randomised, double-blinded, placebo-controlled trial, eligible participants will undergo baseline assessments before being randomised to receive two capsules of placebo twice daily or two capsules of curcumin (corresponding to 200 mg) twice daily for 6 weeks. In the end of the 6-week intervention periods, end-of-trial assessments (similar to baseline assessments) will be performed.

Information meeting:

Prior to any protocol-related procedures, an information meeting at Center for Clinical Metabolic Research, Gentofte Hospital, will be arranged, and subjects will be informed of the possibility of bringing a person of own choice to the visit. During this meeting, a member of the research group will explain the purpose, procedures and possible risks of the study in undisturbed and confidential surroundings. The subject will be informed that if extra time to evaluate participation is needed, a minimum of 24 hours from oral information is given until the consent and sign the informed consent form should be given is acceptable. After obtaining the informed consent, time of screening is planned. The subject will be informed that it is possible to withdraw the written consent at any time prior to or during the study.

Screening visit:

If a person agrees to participate in the study following the information meeting, and oral and written informed consent has been obtained, a screening visit will be planned. The subject will be instructed in a 10 hour overnight fast before screening (including medicine, but water may be consumed until 2 hours before screening). After this fast the subject will meet in the department in the morning. Height and body weight will be measured, medication and medical history will be recorded, blood will be sampled for assessment of plasma/serum concentrations of thyroid-stimulating hormone, creatinine, electrolytes, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), lactate dehydrogenase, alkaline phosphatase, albumin, bilirubin, gamma-glutamyltransferase, viral hepatitis markers, platelet count, ferritin and haemoglobin, and albumin-creatinine ratio in the urine will be measured. A Fibro Scan will be performed. A physical examination will be made including evaluation of blood pressure and pulse rate. Alcohol habits will be evaluated based on The Alcohol Use Disorder Identification Test (AUDIT) questionnaire76,77 and quantification of the weekly amount of alcohol. A magnetic resonance (MR) safety checklist will be completed and a MR information sheet will be given. If all inclusion criteria and none of the exclusion criteria are met, dates for baseline assessments and randomisation visit will be planned within 6 weeks from the screening visit. The subject will be instructed in not to consume curcumin-containing food on a daily basis from screening until end of trial.

Baseline assessments and randomisation visit:

Included subjects will undergo an MRS, which will be scheduled as close as possible to the start of intervention. The subject will meet at the Department of Radiology at Herlev Hospital and be placed in a horizontal position during the scan. During the MRS, a spectroscopy of the liver will be assessed, and an estimation of visceral adipose tissue and subcutaneous adipose tissue will be done. The subject will be placed in a horizontal position during the scan (duration: approximately 30 minutes).

Food and physical activity diary and standardised food intake period: Before start of intervention and during the week before end-of-trial visit, each subject will fill out a three days food and physical activity dairy. The food and physical activity diary will be registered manually by participants, using a questionnaire. The two last days before test days, the participants are requested to have a standardized food intake high in carbohydrates, to get the most valid oral glucose tolerance test (OGTT) response, and the subject will be thoroughly instructed in this.

During the last week before randomisation, the subject is kindly asked to collect a stool sample for the determination of gut bacteria count and subtype. The participant will receive sample kits consisting of cooler bag, freezer packs and stool sample tubes. Stool samples will be collected by the participant at home: Prior to defecation a disposable collector will be placed in the toilet from where stool will be transferred to a tube that immediately is transferred to a transport container and placed at -20°C in the patient's freezer. Prior to transport to Gentofte Hospital, the transport container is transferred to the cooler bag and at arrival at Gentofte Hospital the transport container (with the sample tube) is immediately stored in at -80°C for later analysis. This entails DNA extraction, library preparation, MiSeq 16S rRNA sequencing and microbiota analysis (relative abundance, alpha/beta diversity, link to phenotype of interest).

On the randomisation visit, the subject will meet in the laboratory around 8 a.m. after 10 hours of fast (including medication) and refrainment from tobacco or nicotine supplements use. The subject is allowed to drink water until 8 hours before meeting in department. Furthermore, the subject will be requested to avoid heavy alcohol intake and strenuous exercise two days prior to the visit and instructed to use non-strenuous methods of transportation to the research facility. The following procedures will be conducted:

1. A fasting urine sample will be collected, and the participant is kindly asked to empty the bladder completely. Urine volume will be measured.
2. Measurement of bioimpedance.
3. Fasting blood samples will be collected (genetic markers for NASH, biomarkers of NASH and fibrosis, fibroblast growths factors, triglycerides, cholesterols, liver parameters, haemoglobin A1c, inflammatory markers, adipokines, haemoglobin, creatinine) amounting 22 ml.
4. FibroScan: The subject will be lying in a supine position for approximately 10 minutes during which a probe using shear-waves and ultrasound is applied in the right side of the body below the ribs
5. Measurement of blood pressure, pulse rate, body weight and hip and waist circumference
6. One cannula will be inserted in the cubital vein for collection of blood samples; the forearm from which blood samples are drawn will be wrapped in a heating blanket (42°C) throughout the experiment (for arterialisation of venous blood)
7. Blood samples will be collected according to Table 1 below (total amino acids, gut hormones, glucose, glucagon, insulin, c-peptide, urea, free fatty acids)
8. At time 0 min, the subject will ingest 75 g of water-free glucose dissolved in 300 ml water over a period of 5 minutes
9. At time 0, 30, 60, 90, 120, 150, 180, 210 and 240 min, hunger, satiety, fullness and prospective food consumption will be measured by visual analogue scales (VASs). (see enclosure 5 "VAS").
10. During the last hour (~180min - ~240 min), resting energy expenditure (REE) will be measured in a supine position by indirect calorimetry to determine oxygen consumption (V02) and carbon dioxide production (VC02). A flow-through canopy gas analyser will be used.
11. At time ~240 min the subject will be asked to provide a new urine sample for measurement of urea concentration. The participant is kindly asked to empty the bladder completely. Urine volume will be measured.
12. At time 250 min, the subject will ingest a standardised ad libitum meal consisting of minced meat, pasta, corn, carrots, peppers, cream, salt and pepper (50 energy (E) % carbohydrate, 37 E% fat, 13 E% protein); the subject will be instructed to eat as much as possible until feeling comfortable satiated; the meal should be consumed within a maximum of 30 minutes and by the end of the meal, time spent eating, weight of the meal and the total amount of energy consumed will be noted. Additionally, the participants rated the appearance, smell, taste, off-taste, and overall impression of the ad libitum meal on VAS scores during the ad libitum meal. 10 minutes after termination of the meal consumption, the last questionnaire regarding hunger, satiety, fullness and prospective food consumption will be measured by visual analogue scales.

The interventional period:

The intervention will start soon after randomization visit and first MRS. During the entire intervention period, each subject will fill out a dairy to keep track of any new concomitant medication, compliance and possible adverse events. Each subject will take either two capsules of Meriva® or two placebo capsules each morning and each evening for 42 days (±3 days) with a small glass of water, preferably in relation to a meal. Should the subject forget/miss to take a dose, it can be ingested until 6 hours before the next planned dose. If the subject forgets/misses a dose, and the next planned dose is within the next 6 hours, the dose should be passed, and the subject must note the incident in the diary. The subject is kindly asked to keep the alcohol and smoking habits they might have had before screening and, thus, not to consume more than 21 units of alcohol per week. Furthermore, it is not allowed to consume more than 5 units in one night or to consume curcumin-containing food on a daily basis until end of trial. Mid-way through the intervention period, the subject will receive a phone call from the investigator or other delegated site staff, checking on adverse events, concomitant medication and compliance, and to answer any questions from the subject.

In the last week of intervention, participants are once more requested to fill out questionnaires regarding food intake and physical activity. Starting two days prior to end-of-trial visit, the subject must once more follow two days of standardized food intake.

End-of-trial assessments and visit:

The end-of-trial visit will be scheduled 42±3 days after start of intervention. Within one week prior to the end-of-trial visit, stool sample collection will be scheduled and performed as described above under "Baseline assessments and randomisation visit" and MRS in assessed as close to end-of-trial visit as possible. Procedures during the end-of-trial visit are similar to the ones described above under "Baseline assessments and randomisation visit". Also, during this day, to check for any effect of curcumin intervention, physical examination will be performed by a physician from the research team and additional blood samples (identical with the samples at the screening visit, except viral hepatitis markers) will be collected (which adds another 5 ml blood samples compared to randomisation visit) and albumin-creatinine ratio in the urine will be measured.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30.0 kg/m2
* Haemoglobin ≥7.5 mmol/l
* Written informed consent
* If the subject is known with diet treated diabetes, HbA1c has to be < 48 mmol/mol.
* If the subject is not known diabetes, HbA1c can be <53 mmol/mol

Two of the following four parameters:

* Steatosis on Fibro scan with M-probe or XL-probe (S>=1)
* Waist circumference >94 cm
* HbA1c>48 mmol/mol
* FLI score >60% (see enclosure 2 "FLI score")
* Diagnosis of steatosis on liver biopsy, ultrasound or MR-scan within the last three years and no weight loss or treatment of steatosis since diagnosis. If this inclusion criterion is fulfilled, the BMI criterion written above will not be > 30 kg/m2, but > 27 kg/m2

Exclusion Criteria:

* Use of glucose-lowering drugs, lipid-lowering drugs, warfarin, clopidogrel or non-vitamin K oral anticoagulants
* Treatment with drugs with potential steatogenic side-effects within three months prior to inclusion (e.g. tetracycline, valproic acid, systemic glucocorticoids, amiodarone, tamoxifen and methotrexate)
* Known viral, inherited or alcoholic liver disease, or any other condition known to affect the liver (e.g. coeliac disease, Wilsons disease, cystic fibrosis, alpha-1 anti-trypsin deficiency)
* Positive result of blood test for viral hepatitis markers
* Intake of more than 21 units of alcohol per week, or earlier alcohol abuse
* Frequent use of anti-inflammatory drugs
* Nephropathy (eGFR < 60 ml/min/1.73 m² and/or urine albumin > 20 mg/L)
* In a weight management program, or planning to change life style, alcohol habits or eating habits during the study
* Known allergy to curcumin/turmeric
* Claustrophobia
* Implanted metal objects contraindicative of MRS
* Any condition(s) or clinical or biochemical signs that the investigator think would interfere with trial participation or with the safety of the subject
* Any regular drug treatment that cannot be discontinued for minimum 18 hours

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Curcumin's effect on steatosis | 42 days +/- 3 days
  Percentage of fat in the liver tissue measured by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Curcumin's effect on concentration of total amino acids in plasma | 42 days +/- 3 days
Curcumin's effect on plasma concentration of urea | 42 days +/- 3 days
Curcumin's effect on urin concentration of urea | 42 days +/- 3 days
Curcumin's effect on serum concentration of inflammatory marker interleukin (IL)-1b | 42 days +/- 3 days
Curcumin's effect on serum concentration of inflammatory marker IL-2 | 42 days +/- 3 days
Curcumin's effect on serum concentration of inflammatory marker IL-6 | 42 days +/- 3 days
Curcumin's effect on serum concentration of inflammatory marker IL-10 | 42 days +/- 3 days
Curcumin's effect on serumconcentration of inflammatory marker tumor necrosis factor (TNF)-alpha | 42 days +/- 3 days
Curcumin's effect on plasma concentration of adipokines | 42 days +/- 3 days
Curcumin's effect on plasma concentration of glucagon | 42 days +/- 3 days
Curcumin's effect on plasma concentration of glucagon-like peptide 1 | 42 days +/- 3 days
Curcumin's effect on plasma concentration of glucose-dependent insulinotropic peptide | 42 days +/- 3 days
Curcumin's effect on glucose plasma values during an oral glucose tolerance test for 4 hours | 42 days +/- 3 days
Curcumin's effect on serum c-peptide levels | 42 days +/- 3 days
Curcumin's effect on serum insulin concentration | 42 days +/- 3 days
Curcumin's effect on serum concentration of free fatty acids | 42 days +/- 3 days
Curcumin's effect on liver insulin resistance | 42 days +/- 3 days
Curcumin's effect on body weight in kilograms | 42 days +/- 3 days
Curcumin's effect on BMI (kg/m^2) | 42 days +/- 3 days
Curcumin's effect on waist circumference (cm) | 42 days +/- 3 days
Curcumin's effect on waist-hip ratio | 42 days +/- 3 days
Curcumin's effect on systolic blood pressure (mmHg) | 42 days +/- 3 days
Curcumin's effect on diastolic blood pressure (mmHg) | 42 days +/- 3 days
Curcumin's effect on transient elastography liver stiffness measurements (kPa) | 42 days +/- 3 days
  Evaluated with FibroScan
Curcumin's effect on transient elastography controlled attenuation parameter (CAP) value (dB/m) | 42 days +/- 3 days
  Evaluated with FibroScan
Curcumin's effect on gut microbiota (relative abundance) | 42 days +/- 3 days
Curcumin's effect on gut microbiota (alpha/beta diversity) | 42 days +/- 3 days
Curcumin's effect on gut microbiota (link to phenotype of interest) | 42 days +/- 3 days
Curcumin's effect on visceral fat (cm) | 42 days +/- 3 days
  Evaluated by MR-spectroscopy
Curcumin's effect on subcutaneous fat (cm) | 42 days +/- 3 days
  Evaluated by MR-spectroscopy
Curcumin's effect on muscle percentage | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on fatt mass | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on fat percentage | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on fat-free mass | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on fat-free mass percentage | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on total body water | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on body water percentage | 42 days +/- 3 days
  Evaluated by bioimpedance measurement
Curcumin's effect on prospective food consumption | 42 days +/- 3 days
  Evaluated by questionnaires during the OGTT on the experimental days
Curcumin's effect on food consumption | 42 days +/- 3 days
  Evaluated by how many grams of standardised meal the subject eats at an ad libitum meal
Curcumin's effect on calory balance | 42 days +/- 3 days
  Evaluated by a questionnaire participants fill out on 3 consecutive days
Curcumin's effect on plasma concentration of cholesterol | 42 days +/- 3 days
Curcumin's effect on plasma concentration of alanine aminotransferase | 42 days +/- 3 days
Curcumin's effect on plasma concentration of aspartate aminotransferase | 42 days +/- 3 days
Genetic risk markers for development of NASH | On both test days

CONTACTS AND LOCATIONS:
Overall Officials: Pernille H Hellmann, MD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No